CLINICAL TRIAL: NCT05641818
Title: Challenges in Achieving Adequate Vitamin D Status in the Adult Population - Part 3: Screening Tool for Identification of Subjects at Risk for Suboptimal Vitamin D Status
Brief Title: Challenges in Achieving Adequate Vitamin D Status in the Adult Population - Part 3 (VITAD/3)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: National Institute of Public Health, Slovenia (Other Government); VIST - Faculty of Applied Sciences (Other); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Other Study IDs: VITAD-01-2018 Part 3
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Vitamin D Serum Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Screening tool for vitamin D deficiency — (1) Determination of 25(OH) Vitamin D3 in human serum samples and (2) Question based screening tool with personal (age, gender,...), lifestyle (e.g. sun exposure, outdoor activity) and dietary factors that affect the status of vitamin D in the human body.

SUMMARY:
Validation of a screening tool for identification of subjects at risk for suboptimal vitamin D status. Developed questionnaire-based screening tool will be used on subjects with various risks for vitamin D deficiency, and compared with 25-OH-vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed consent form (ICF),
* Age between 18 and 65 years at the time of the signature of Informed consent form (ICF),
* Did not change use of vitamin D conatining drugs/supplements for last 6 weeks
* Willingness to follow all study procedures

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Change in use of food supplements containing Vitamin D in last 6 weeks
* Acute ilness
* Mental incapacity that precludes adequate understanding or cooperation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult users and non-users of vitamin D drugs and food supplements living in Slovenia. Participants invited from the database at Nutrition Institute.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference between vitamin D status (deficiency) assessed by two different methods | 1 year
  Vitamin D serum level will be measured for assessment of Vitamin D status. Risk for vitamin D deficiency will be assessed using questionaire-based screening tool. Two methods will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, PhD, Study Chair — Institut za nutricionistiko; Katja Žmitek, PhD, Principal Investigator — VIST - Faculty of Applied Sciences
Locations (1):
- Nutrition Institute, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet